CLINICAL TRIAL: NCT00450918
Title: Longitudinal Study of Primary Ciliary Dyskinesia: Participants 5-18 Years of Age
Brief Title: Evaluating Progression of and Diagnostic Tools for Primary Ciliary Dyskinesia in Children and Adolescents
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Office of Rare Diseases (ORD) (NIH); National Center for Research Resources (NCRR) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 05-2997; U54HL096458 (NIH); RDCRN 5901 (Other: UNC)
Record Dates: First submitted 2007-03-20; First posted 2007-03-22 (Estimated); Last update posted 2019-10-07 (Actual); Status verified 2019-10

CONDITIONS: Primary Ciliary Dyskinesia
Keywords: Kartagener Syndrome
MeSH Terms: conditions — Ciliary Motility Disorders; Kartagener Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Mucociliary clearance, in which mucus secretions are cleared from the breathing airways, is the primary defense mechanism for the lungs. Inhaled particles, including microbes that can cause infections, are normally entrapped in mucus on the airway surfaces and then cleared out by the coordinated action of tiny hair-like structures called cilia. Individuals with primary ciliary dyskinesia (PCD) have defective mucociliary clearance, which in turn leads to lung infections and disease. The purpose of this study is to determine how lung disease progresses over time in children and adolescents with PCD.

DETAILED DESCRIPTION:
PCD is a rare genetic disorder in which impaired mucus clearance commonly results in chronic cough and infections in the airways, sinuses, and middle ears. Long lasting airway infection ultimately leads to structural damage to the airways, known as bronchiectasis, and, in turn, loss of lung function. While PCD shares some similarities with the disease cystic fibrosis, it is important to distinguish PCD from cystic fibrosis. In particular, the age of onset and progression of PCD's clinical lung disease, including timing of specific microbial pathogen infections and bronchiectasis, remain poorly defined. The purpose of this study is to determine how lung disease progresses over time in children and adolescents with PCD. Specific attention will be directed toward determining whether certain factors play a role in lung disease progression. The study will also evaluate diagnostic tools and quality of life among individuals with PCD. Filling these gaps of knowledge may help to improve the clinical management of PCD in the future.

This longitudinal study will last 5 years. There will be a total of 5 study visits, and these visits will occur yearly. Each study visit will last 3 to 4 hours. All study visits will include a medical history review; physical exam; height, weight, and vital sign measurements; sampling of respiratory fluids and mucus; lung function tests; and questionnaires. The initial visit may also include using a probe to measure nasal nitric oxide levels and blood collection for genetic testing. Study visits 1, 3, and 5 will also include blood collection for pregnancy testing and a high resolution computed tomography (HRCT) scan of the chest to image the lungs. At the end of each month, participants will report any use of oral, inhaled, or intravenous antibiotics.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of PCD or probable PCD. More information about the criteria for a PCD diagnosis can be found in the protocol.
* Parent or guardian willing to provide informed consent

Exclusion Criteria:

* Inability to attend follow-up appointments
* Previously received lung transplant
* Any disease that may have significant impact on lung function (e.g., severe congenital heart disease, severe scoliosis), respiratory infections (e.g., AIDS), or overall health status (e.g., cancer, end-stage kidney disease)
* Pregnant or breastfeeding

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children and adolescents with primary ciliary dyskinesia
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2006-08; Primary Completion 2019-08 (Actual); Study Completion 2019-08 (Actual)

PRIMARY OUTCOMES:
Spirometry Measures | Measured yearly for 5 years
HRCT scan of the chest to image lungs | At visits 1, 3, and 5

CONTACTS AND LOCATIONS:
Overall Officials: Margaret W Leigh, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (5):
- United States (4):
  - The Children's Hospital, Denver, Colorado
  - Washington University, St Louis, Missouri
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Children's Hospital and Regional Medical Center, Seattle, Washington
- The Hospital for Sick Children, Toronto, Ontario, Canada

REFERENCES:
- [Background] Corbelli R, Bringolf-Isler B, Amacher A, Sasse B, Spycher M, Hammer J. Nasal nitric oxide measurements to screen children for primary ciliary dyskinesia. Chest. 2004 Oct;126(4):1054-9. doi: 10.1378/chest.126.4.1054. PMID 15486363
- [Background] Hossain T, Kappelman MD, Perez-Atayde AR, Young GJ, Huttner KM, Christou H. Primary ciliary dyskinesia as a cause of neonatal respiratory distress: implications for the neonatologist. J Perinatol. 2003 Dec;23(8):684-7. doi: 10.1038/sj.jp.7210987. PMID 14647169
- [Background] Noone PG, Leigh MW, Sannuti A, Minnix SL, Carson JL, Hazucha M, Zariwala MA, Knowles MR. Primary ciliary dyskinesia: diagnostic and phenotypic features. Am J Respir Crit Care Med. 2004 Feb 15;169(4):459-67. doi: 10.1164/rccm.200303-365OC. Epub 2003 Dec 4. PMID 14656747
- [Background] Fliegauf M, Olbrich H, Horvath J, Wildhaber JH, Zariwala MA, Kennedy M, Knowles MR, Omran H. Mislocalization of DNAH5 and DNAH9 in respiratory cells from patients with primary ciliary dyskinesia. Am J Respir Crit Care Med. 2005 Jun 15;171(12):1343-9. doi: 10.1164/rccm.200411-1583OC. Epub 2005 Mar 4. PMID 15750039
- [Background] Horvath J, Fliegauf M, Olbrich H, Kispert A, King SM, Mitchison H, Zariwala MA, Knowles MR, Sudbrak R, Fekete G, Neesen J, Reinhardt R, Omran H. Identification and analysis of axonemal dynein light chain 1 in primary ciliary dyskinesia patients. Am J Respir Cell Mol Biol. 2005 Jul;33(1):41-7. doi: 10.1165/rcmb.2004-0335OC. Epub 2005 Apr 21. PMID 15845866
- [Background] Zariwala MA, Leigh MW, Ceppa F, Kennedy MP, Noone PG, Carson JL, Hazucha MJ, Lori A, Horvath J, Olbrich H, Loges NT, Bridoux AM, Pennarun G, Duriez B, Escudier E, Mitchison HM, Chodhari R, Chung EM, Morgan LC, de Iongh RU, Rutland J, Pradal U, Omran H, Amselem S, Knowles MR. Mutations of DNAI1 in primary ciliary dyskinesia: evidence of founder effect in a common mutation. Am J Respir Crit Care Med. 2006 Oct 15;174(8):858-66. doi: 10.1164/rccm.200603-370OC. Epub 2006 Jul 20. PMID 16858015
- [Background] Kennedy MP, Noone PG, Carson J, Molina PL, Ghio A, Zariwala MA, Minnix SL, Knowles MR. Calcium stone lithoptysis in primary ciliary dyskinesia. Respir Med. 2007 Jan;101(1):76-83. doi: 10.1016/j.rmed.2006.04.007. Epub 2006 Jun 6. PMID 16757159
- [Background] Hornef N, Olbrich H, Horvath J, Zariwala MA, Fliegauf M, Loges NT, Wildhaber J, Noone PG, Kennedy M, Antonarakis SE, Blouin JL, Bartoloni L, Nusslein T, Ahrens P, Griese M, Kuhl H, Sudbrak R, Knowles MR, Reinhardt R, Omran H. DNAH5 mutations are a common cause of primary ciliary dyskinesia with outer dynein arm defects. Am J Respir Crit Care Med. 2006 Jul 15;174(2):120-6. doi: 10.1164/rccm.200601-084OC. Epub 2006 Apr 20. PMID 16627867
- [Background] Kennedy MP, Ostrowski LE. Primary ciliary dyskinesia and upper airway diseases. Curr Allergy Asthma Rep. 2006 Nov;6(6):513-7. doi: 10.1007/s11882-006-0030-7. PMID 17026878
- [Background] Ferkol T, Leigh M. Primary ciliary dyskinesia and newborn respiratory distress. Semin Perinatol. 2006 Dec;30(6):335-40. doi: 10.1053/j.semperi.2005.11.001. PMID 17142159
- [Background] Zariwala MA, Despotes KA, Davis SD. Primary Ciliary Dyskinesia. 2007 Jan 24 [updated 2025 May 22]. In: Adam MP, Bick S, Mirzaa GM, Pagon RA, Wallace SE, Amemiya A, editors. GeneReviews(R) [Internet]. Seattle (WA): University of Washington, Seattle; 1993-2026. Available from http://www.ncbi.nlm.nih.gov/books/NBK1122/ PMID 20301301
- [Background] Kennedy MP, Noone PG, Leigh MW, Zariwala MA, Minnix SL, Knowles MR, Molina PL. High-resolution CT of patients with primary ciliary dyskinesia. AJR Am J Roentgenol. 2007 May;188(5):1232-8. doi: 10.2214/AJR.06.0965. PMID 17449765
- [Background] Zariwala MA, Knowles MR, Omran H. Genetic defects in ciliary structure and function. Annu Rev Physiol. 2007;69:423-50. doi: 10.1146/annurev.physiol.69.040705.141301. PMID 17059358
- [Background] Morillas HN, Zariwala M, Knowles MR. Genetic causes of bronchiectasis: primary ciliary dyskinesia. Respiration. 2007;74(3):252-63. doi: 10.1159/000101783. PMID 17534128
- [Background] Kennedy MP, Omran H, Leigh MW, Dell S, Morgan L, Molina PL, Robinson BV, Minnix SL, Olbrich H, Severin T, Ahrens P, Lange L, Morillas HN, Noone PG, Zariwala MA, Knowles MR. Congenital heart disease and other heterotaxic defects in a large cohort of patients with primary ciliary dyskinesia. Circulation. 2007 Jun 5;115(22):2814-21. doi: 10.1161/CIRCULATIONAHA.106.649038. Epub 2007 May 21. PMID 17515466
- [Background] Loges NT, Olbrich H, Becker-Heck A, Haffner K, Heer A, Reinhard C, Schmidts M, Kispert A, Zariwala MA, Leigh MW, Knowles MR, Zentgraf H, Seithe H, Nurnberg G, Nurnberg P, Reinhardt R, Omran H. Deletions and point mutations of LRRC50 cause primary ciliary dyskinesia due to dynein arm defects. Am J Hum Genet. 2009 Dec;85(6):883-9. doi: 10.1016/j.ajhg.2009.10.018. PMID 19944400
- [Background] Leigh MW, Pittman JE, Carson JL, Ferkol TW, Dell SD, Davis SD, Knowles MR, Zariwala MA. Clinical and genetic aspects of primary ciliary dyskinesia/Kartagener syndrome. Genet Med. 2009 Jul;11(7):473-87. doi: 10.1097/GIM.0b013e3181a53562. PMID 19606528
- [Background] Lie H, Zariwala MA, Helms C, Bowcock AM, Carson JL, Brown DE 3rd, Hazucha MJ, Forsen J, Molter D, Knowles MR, Leigh MW, Ferkol TW. Primary ciliary dyskinesia in Amish communities. J Pediatr. 2010 Jun;156(6):1023-1025. doi: 10.1016/j.jpeds.2010.01.054. Epub 2010 Mar 29. PMID 20350728
- [Background] Griggs RC, Batshaw M, Dunkle M, Gopal-Srivastava R, Kaye E, Krischer J, Nguyen T, Paulus K, Merkel PA; Rare Diseases Clinical Research Network. Clinical research for rare disease: opportunities, challenges, and solutions. Mol Genet Metab. 2009 Jan;96(1):20-6. doi: 10.1016/j.ymgme.2008.10.003. Epub 2008 Nov 13. PMID 19013090
- [Background] Olin JT, Burns K, Carson JL, Metjian H, Atkinson JJ, Davis SD, Dell SD, Ferkol TW, Milla CE, Olivier KN, Rosenfeld M, Baker B, Leigh MW, Knowles MR, Sagel SD; Genetic Disorders of Mucociliary Clearance Consortium. Diagnostic yield of nasal scrape biopsies in primary ciliary dyskinesia: a multicenter experience. Pediatr Pulmonol. 2011 May;46(5):483-8. doi: 10.1002/ppul.21402. Epub 2011 Jan 31. PMID 21284095
- [Background] Zariwala MA, Omran H, Ferkol TW. The emerging genetics of primary ciliary dyskinesia. Proc Am Thorac Soc. 2011 Sep;8(5):430-3. doi: 10.1513/pats.201103-023SD. PMID 21926394
- [Background] Leigh MW, O'Callaghan C, Knowles MR. The challenges of diagnosing primary ciliary dyskinesia. Proc Am Thorac Soc. 2011 Sep;8(5):434-7. doi: 10.1513/pats.201103-028SD. PMID 21926395
- [Background] Davis SD, Knowles M, Leigh M. Introduction: primary ciliary dyskinesia and overlapping syndromes. Proc Am Thorac Soc. 2011 Sep;8(5):421-2. doi: 10.1513/pats.201103-026SD. No abstract available. PMID 21926392
- [Background] Ostrowski LE, Dutcher SK, Lo CW. Cilia and models for studying structure and function. Proc Am Thorac Soc. 2011 Sep;8(5):423-9. doi: 10.1513/pats.201103-027SD. PMID 21926393
- [Background] Mateos-Corral D, Coombs R, Grasemann H, Ratjen F, Dell SD. Diagnostic value of nasal nitric oxide measured with non-velum closure techniques for children with primary ciliary dyskinesia. J Pediatr. 2011 Sep;159(3):420-4. doi: 10.1016/j.jpeds.2011.03.007. Epub 2011 Apr 22. PMID 21514598
- [Background] Knowles MR, Leigh MW, Carson JL, Davis SD, Dell SD, Ferkol TW, Olivier KN, Sagel SD, Rosenfeld M, Burns KA, Minnix SL, Armstrong MC, Lori A, Hazucha MJ, Loges NT, Olbrich H, Becker-Heck A, Schmidts M, Werner C, Omran H, Zariwala MA; Genetic Disorders of Mucociliary Clearance Consortium. Mutations of DNAH11 in patients with primary ciliary dyskinesia with normal ciliary ultrastructure. Thorax. 2012 May;67(5):433-41. doi: 10.1136/thoraxjnl-2011-200301. Epub 2011 Dec 18. PMID 22184204
- [Background] Stillwell PC, Wartchow EP, Sagel SD. Primary Ciliary Dyskinesia in Children: A Review for Pediatricians, Allergists, and Pediatric Pulmonologists. Pediatr Allergy Immunol Pulmonol. 2011 Dec;24(4):191-196. doi: 10.1089/ped.2011.0099. PMID 22276227
- [Background] Knowles MR, Leigh MW, Zariwala MA. Cutting edge genetic studies in primary ciliary dyskinesia. Thorax. 2012 May;67(5):464; author reply 464. doi: 10.1136/thoraxjnl-2012-201609. Epub 2012 Feb 10. No abstract available. PMID 22328589
- [Background] Horani A, Druley TE, Zariwala MA, Patel AC, Levinson BT, Van Arendonk LG, Thornton KC, Giacalone JC, Albee AJ, Wilson KS, Turner EH, Nickerson DA, Shendure J, Bayly PV, Leigh MW, Knowles MR, Brody SL, Dutcher SK, Ferkol TW. Whole-exome capture and sequencing identifies HEATR2 mutation as a cause of primary ciliary dyskinesia. Am J Hum Genet. 2012 Oct 5;91(4):685-93. doi: 10.1016/j.ajhg.2012.08.022. PMID 23040496
- [Background] Ferkol TW, Leigh MW. Ciliopathies: the central role of cilia in a spectrum of pediatric disorders. J Pediatr. 2012 Mar;160(3):366-71. doi: 10.1016/j.jpeds.2011.11.024. Epub 2011 Dec 16. No abstract available. PMID 22177992
- [Background] Nakhleh N, Francis R, Giese RA, Tian X, Li Y, Zariwala MA, Yagi H, Khalifa O, Kureshi S, Chatterjee B, Sabol SL, Swisher M, Connelly PS, Daniels MP, Srinivasan A, Kuehl K, Kravitz N, Burns K, Sami I, Omran H, Barmada M, Olivier K, Chawla KK, Leigh M, Jonas R, Knowles M, Leatherbury L, Lo CW. High prevalence of respiratory ciliary dysfunction in congenital heart disease patients with heterotaxy. Circulation. 2012 May 8;125(18):2232-42. doi: 10.1161/CIRCULATIONAHA.111.079780. Epub 2012 Apr 12. PMID 22499950
- [Background] Antony D, Becker-Heck A, Zariwala MA, Schmidts M, Onoufriadis A, Forouhan M, Wilson R, Taylor-Cox T, Dewar A, Jackson C, Goggin P, Loges NT, Olbrich H, Jaspers M, Jorissen M, Leigh MW, Wolf WE, Daniels ML, Noone PG, Ferkol TW, Sagel SD, Rosenfeld M, Rutman A, Dixit A, O'Callaghan C, Lucas JS, Hogg C, Scambler PJ, Emes RD; Uk10k; Chung EM, Shoemark A, Knowles MR, Omran H, Mitchison HM. Mutations in CCDC39 and CCDC40 are the major cause of primary ciliary dyskinesia with axonemal disorganization and absent inner dynein arms. Hum Mutat. 2013 Mar;34(3):462-72. doi: 10.1002/humu.22261. Epub 2013 Feb 11. PMID 23255504
- [Background] Sears PR, Thompson K, Knowles MR, Davis CW. Human airway ciliary dynamics. Am J Physiol Lung Cell Mol Physiol. 2013 Feb 1;304(3):L170-83. doi: 10.1152/ajplung.00105.2012. Epub 2012 Nov 9. PMID 23144323
- [Background] Knowles MR, Leigh MW, Ostrowski LE, Huang L, Carson JL, Hazucha MJ, Yin W, Berg JS, Davis SD, Dell SD, Ferkol TW, Rosenfeld M, Sagel SD, Milla CE, Olivier KN, Turner EH, Lewis AP, Bamshad MJ, Nickerson DA, Shendure J, Zariwala MA; Genetic Disorders of Mucociliary Clearance Consortium. Exome sequencing identifies mutations in CCDC114 as a cause of primary ciliary dyskinesia. Am J Hum Genet. 2013 Jan 10;92(1):99-106. doi: 10.1016/j.ajhg.2012.11.003. Epub 2012 Dec 20. PMID 23261302
- [Background] Ferkol TW, Puffenberger EG, Lie H, Helms C, Strauss KA, Bowcock A, Carson JL, Hazucha M, Morton DH, Patel AC, Leigh MW, Knowles MR, Zariwala MA. Primary ciliary dyskinesia-causing mutations in Amish and Mennonite communities. J Pediatr. 2013 Aug;163(2):383-7. doi: 10.1016/j.jpeds.2013.01.061. Epub 2013 Mar 7. PMID 23477994